# UC Davis and UC Davis Health Consent to Participate in Research

**Title of study:** Using an AI mobile application to promote healthy eating **Principal Investigator:** Lauren Au, PhD RDN

**Date approved: 06/04/2025** 

If you agree to take part, you will be given a copy of this document.

Do not write below this line. For IRB stamp and version date only.

### **Introduction and Purpose**

You are invited to be part of a research study. The goal of this study is to test how well a mobile app called PlantVillage Food works for students at UC Davis.

The risks of this research are minimal. Some of the questions might make you feel uncomfortable or upset. You do not have to answer any of the questions you do not want to answer.

### **Validation Study**

If you join this study, you will visit the dining commons on three different days.

- Day 1:
  - o You'll learn about the study, sign a consent form, and receive training.
  - o You'll fill out a survey (about 20 minutes total).
  - o You'll also learn how to install and use the app (about 20–30 minutes).
  - The whole visit should take 40–50 minutes.
- Days 2 & 3:
  - o On two separate days, you'll use the app to record the foods you eat.
  - o Research staff will weigh your food before and after you eat.

#### **Timeline**

Happens over 3 days during Fall 2025. Expect about 1 hour for the first visit and 5-7 total hours for the other two days.

#### What to Know Before You Join

- The study uses photos of your food, but no personal information about you will be shared.
- Your information will be kept private and only approved researchers will be able to see it.
- You don't have to join. If you do join, you can stop at any time without losing any UC Davis benefits.
- If you want your data removed from the study later, just contact the research team.

#### **Benefits**

You won't get any personal health benefits from joining. But the research could help us learn more about how mobile apps and AI can support healthy eating.

Joining or leaving the study will not affect your status as a UC Davis student.

## **Confidentiality**

As with all research, there is a chance that confidentiality could be compromised; however, we are taking precautions to minimize this risk. Your responses to the survey will not include information that identifies you. However, individuals from UC Davis who oversee research may access your data during audits or other monitoring activities.

To minimize the risks of breaching confidentiality, we will remove any identification that links you to your data. Additionally, the data will be coded and stored in a password-protected Box folder accessible only by the PI and project manager.

We will use your information to conduct this study. Leftover data collected for this research may also be used for future research studies. We will not share any personally

Do not write below this line. For IRB stamp and version date only.

identifiable information. Our goal is to make more research possible. These studies may be done by researchers at this institution or other institutions, including commercial entities. Data may be placed in one or more external scientific databases for access and use. We will not ask you for additional permission to share de-identified information.

## **Rights**

Taking part in research is completely voluntary. You are free to decline to take part in the project. You can decline to answer any questions, and you can stop taking part in the project at any time. Whether or not you choose to take part, answer any question, or stop taking part in the project, there will be no penalty to you or loss of benefits to which you are otherwise entitled. We will use your information to conduct this study. Data collected for this research may also be used for future research studies. We will not share any personally identifiable information. Our goal is to make more research possible. These studies may be done by researchers at this institution or other institutions, including commercial entities. Data may be placed in one or more external scientific databases for access and use. We will not ask you for additional permission to share deidentified

### Compensation

If you join, you can earn up to:

- Up to \$50 in gift cards:
  - o \$15 after Day 2
  - o \$35 after Day 3

#### **Ouestions**

If you have any questions about this research, or you believe that you've been injured or harmed as a participant in this research, please contact the investigator at <a href="mailto:leau@ucdavis.edu">leau@ucdavis.edu</a>.

If you have any questions about your rights or treatment as a research participant in this study, please contact the UC Davis, Institutional Review Board by phone: 916-703-9158 or by email: HS-IRBEducation@ucdavis.edu.

Do not write below this line. For IRB stamp and version date only.